CLINICAL TRIAL: NCT07372365
Title: Orelabrutinib as Consolidation and Maintenance Therapy in Treatment-Naïve Marginal Zone Lymphoma: A Study of Efficacy and Safety.
Brief Title: Orelabrutinib as Consolidation and Maintenance Therapy in Treatment-Naïve MZL.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025808
Record Dates: First submitted 2025-12-22; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib Consolidation and Maintenance Therapy in Marginal Zone Lymphoma (Experimental): Eligible subjects will receive R-CHOP regimen (with a 21-day cycle). After 3 cycles of treatment, the efficacy will be assessed. Subjects with disease progression or those who do not achieve partial remission (PR) after treatment will discontinue treatment. The remaining subjects will continue to receive 3 cycles of OR regimen for consolidation therapy. After 6 cycles, efficacy will be assessed again. Subjects assessed as complete remission (CR) or PR will enter the orelabrutinib maintenance treatment phase for a total of 2 years, until completion of the protocol treatment, disease progression, or unacceptable toxicity (whichever occurs first).
  Interventions: Drug: Orelabrutinib Consolidation and Maintenance Therapy

INTERVENTIONS:
Drug: Orelabrutinib Consolidation and Maintenance Therapy — Eligible subjects will receive R-CHOP regimen (with a 21-day cycle). After 3 cycles of treatment, the efficacy will be assessed. Subjects with disease progression or those who do not achieve partial remission (PR) after treatment will discontinue treatment. The remaining subjects will continue to receive 3 cycles of OR regimen for consolidation therapy. After 6 cycles, efficacy will be assessed again. Subjects assessed as complete remission (CR) or PR will enter the orelabrutinib maintenance treatment phase for a total of 2 years, until completion of the protocol treatment, disease progression, or unacceptable toxicity (whichever occurs first).

SUMMARY:
This study aims to explore a new treatment approach for patients with treatment-naive Marginal Zone Lymphoma (MZL). MZL is a type of slow-growing lymphoma that often affects older adults. The current standard treatment involves chemotherapy, but it can have significant side effects and may not always provide long-term benefits. This study investigates a treatment strategy that combines a limited course of chemotherapy (R-CHOP) followed by consolidation and maintenance therapy with a targeted drug called Orelabrutinib.

Patients will undergo a series of tests to determine eligibility for the study. These tests include blood work, imaging studies, and assessments of overall health. Eligible participants will receive a standard chemotherapy regimen called R-CHOP for three cycles. After this, the response to treatment will be evaluated. Participants who show a good response will then receive three cycles of consolidation therapy with Orelabrutinib and Rituximab (OR). Those who continue to respond well will enter a maintenance phase with Orelabrutinib for up to two years. Throughout the study, participants will be closely monitored for treatment response and any side effects. Regular check-ups, blood tests, and imaging studies will be conducted to assess the effectiveness and safety of the treatment.

This study is an important step towards finding better treatment options for MZL patients. It is hoped that through this research, the quality of life and outcomes for those affected by this disease can be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20-positive marginal zone lymphoma (MZL) that has not received systemic therapy.
2. MZL that has progressed or relapsed after prior local therapy (local therapy includes surgery, radiotherapy, Helicobacter pylori eradication, and hepatitis C treatment) or is not amenable to local therapy.
3. Age ≥18 years.
4. Presence of an indication for treatment as determined by the investigator or patient's willingness to receive treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.
6. Adequate organ function as defined below:

   * Hematology: Hemoglobin (HB) ≥60 g/L, platelets (PLT) ≥50×10⁹/L, neutrophils (NE) ≥1.0×10⁹/L (Note: Subjects with cytopenia due to lymphoma bone marrow involvement are not restricted by this criterion).
   * Cardiac: Left ventricular ejection fraction (LVEF) ≥50% as determined by echocardiogram.
   * Renal: Creatinine ≤1.5×upper limit of normal (ULN) or creatinine clearance ≥30 ml/min.
   * Hepatic: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN.
7. Women of childbearing potential must have a negative pregnancy test. Both male and female patients must agree to use effective contraception during the treatment period and for 2 years thereafter.
8. Life expectancy of more than 3 months.
9. Voluntary provision of written informed consent.

Exclusion Criteria:

1. Underwent major surgery or severe trauma within 2 weeks prior to enrollment, or has not yet recovered from significant adverse effects.
2. Has other malignancies currently or within the past 3 years, excluding those that have been cured (such as basal or squamous cell carcinoma of the skin, superficial bladder cancer, prostatic intraepithelial neoplasia, and cervical carcinoma in situ).
3. Has a history of stroke or intracranial hemorrhage within the past 3 months.
4. Requires anticoagulation with warfarin or equivalent vitamin K antagonist.
5. Has evidence of any comorbidities or medical conditions that may interfere with the conduct of the study or place the patient at significant risk, including but not limited to severe cardiovascular disease (e.g., New York Heart Association class III or IV heart disease, myocardial infarction within the past 6 months, unstable arrhythmia, or unstable angina) and/or severe pulmonary disease (e.g., severe obstructive pulmonary disease and a history of symptomatic bronchospasm).
6. Is infected with human immunodeficiency virus, or has uncontrollable active hepatitis C virus or hepatitis B virus infection.
7. Has uncontrollable active infection.
8. Is pregnant or breastfeeding.
9. Has any life-threatening disease, medical condition, or organ dysfunction that may jeopardize the safety of the patient, as determined by the investigator.
10. Has any condition that may interfere with the absorption or metabolism of orelabrutinib or place the study results at unnecessary risk.
11. Has central nervous system involvement by marginal zone lymphoma or evidence of disease transformation.
12. Has any condition that the investigator judges may interfere with the patient's full participation in the study; any condition that poses significant risk to the patient; or any condition that may interfere with the interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate after 6 treatment cycles | Efficacy will be assessed at the end of the combined induction and consolidation therapy (6 cycles in total). Each treatment cycle is 21 days.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From the first dose of study treatment until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months.
Overall survival（OS） | From the first dose of study treatment until the date of death from any cause, assessed up to 60 months.
Overall Response Rate (ORR) after 6 treatment cycles | Efficacy will be assessed at the end of the combined induction and consolidation therapy (6 cycles in total). Each treatment cycle is 21 days.
Adverse events | From the first dose of study treatment until 30 days after the last dose, or until the start of new anti-cancer therapy, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China